CLINICAL TRIAL: NCT00002897
Title: RANDOMIZED STUDY OF PREOPERATIVE CHEMOTHERAPY VERSUS SURGERY ALONE IN ESOPHAGUS CANCER
Brief Title: Surgery With or Without Chemotherapy in Treating Patients With Stage II or Stage III Cancer of the Esophagus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065226; CNR-012809; EU-96038
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-05

CONDITIONS: Esophageal Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not known whether chemotherapy before surgery is more effective than surgery alone in treating cancer of the esophagus.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without chemotherapy in treating patients with stage II or stage III cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare resectability and survival in patients with stage II/III esophageal cancer treated with neoadjuvant cisplatin/fluorouracil vs. surgery alone.

OUTLINE: This is a randomized study. Patients are randomized to one of two groups. The first group receives cisplatin and fluorouracil every 4 weeks for 3 courses followed by esophagectomy and regional lymphadenectomy. The second group undergoes esophagectomy and regional lymphadenectomy alone. All patients are followed for survival.

PROJECTED ACCRUAL: A total of 240 patients will be entered over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed esophageal squamous cell cancer that is stage T2-3 Nx M0

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: WHO 0-2 Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No second malignancy within 5 years except: Basal cell skin carcinoma Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: No prior chemotherapy or radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 1992-07; Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ermanno Ancona, MD, Study Chair — Azienda Ospedaliera di Padova
Locations (1):
- University of Padua, Padua, Italy

REFERENCES:
- [Result] Ancona E, Ruol A, Santi S, Merigliano S, Sileni VC, Koussis H, Zaninotto G, Bonavina L, Peracchia A. Only pathologic complete response to neoadjuvant chemotherapy improves significantly the long term survival of patients with resectable esophageal squamous cell carcinoma: final report of a randomized, controlled trial of preoperative chemotherapy versus surgery alone. Cancer. 2001 Jun 1;91(11):2165-74. PMID 11391598
- [Result] Ancona E, Ruol A, Santi S, et al.: Major response to neoadjuvant chemotherapy leads to improved long-term survival in potentially resectable (T2-3, any N, M0) esophageal squamous cell carcinoma. Final report of a randomized trial of neoadjuvant chemotherapy versus surgery alone. [Abstract] Proceedings of the European Surgical Association 7th annual meeting, Amsterdam, April 14-15, 2000.